CLINICAL TRIAL: NCT04403152
Title: Five Days of Intensive Postoperative Rehabilitation is Superior Than Mobilization in Improving Length of Hospitalization and Outcome of Patients Having Scoliosis Surgery: A Randomized Controlled Trial
Brief Title: Postoperative Rehabilitation or Mobilization After Scoliosis Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Zilan Bazancir Apaydın, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017/53
Record Dates: First submitted 2020-05-21; First posted 2020-05-27 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Scoliosis Idiopathic; Scoliosis; Adolescence
Keywords: rehabilitation; post-operative; early ambulation; posterior fusion surgery
MeSH Terms: conditions — Scoliosis | interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Masking Description: The patients and the researcher who were responsible for the analyzing of the data were blinded to the randomization results.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehabilitation group (Experimental): This is the study group in whom post-operative rehabilitation was provided for 5 days.
  Interventions: Other: Post-operative rehabilitation
- Mobilization group (Active Comparator): This is the control group in whom post-operative mobilization was provided for 5 days.
  Interventions: Other: Post-operative mobilization

INTERVENTIONS:
Other: Post-operative rehabilitation — Patients received the exercises programme for five days, 30 minutes, two times per day with supervision by a physical therapist.
  Other Names: rehabilitation
  Arms: Rehabilitation group
Other: Post-operative mobilization — Patients received usual mobilization programme for 2-5 minutes, two times per day the five days with supervision by a physical therapist.
  Other Names: mobilization
  Arms: Mobilization group

SUMMARY:
Scoliosis surgery is a major surgery associated with postoperative pain, loss of physical function and pulmonary dysfunction in adolescent idiopathic scoliosis patients (AIS).Despite the advanced, various medical treatment methods of pain applied in the postoperative period, the mean period of hospitalization is 5 to 7 days. The increasing health expenditures over the years have brought along the need for rehabilitation programs conducted in the early term. Although early mobilization has been accepted as a rule of thumb by spinal surgeons in preventing the performance loss and reducing the causes of morbidity in recent years, the investigators could not find any research on postoperative rehabilitation implemented on patients under the supervision of a physiotherapist, following scoliosis surgery. The aim of this study was to compare effect of five days of intensive postoperative rehabilitation and mobilization on length of hospitalization and outcome in patients having scoliosis surgery.

DETAILED DESCRIPTION:
Following spinal surgeries, patients experienced deep somatic pain and severe reflex spasms of the muscles located in the surgical site. In addition, pulmonary dysfunction could develop due to reduced flexibility of the spine and mobility of the ribs. It is a known fact that cardiopulmonary functions in adolescent idiopathic scoliosis patients may not recover even two years after surgery. After fusion surgeries in patients with scoliosis have shown that the static and dynamic postural control were impaired and that the postural control could recover one year after the surgery. The increasing health expenditures over the years have brought along the need for rehabilitation programs conducted in the early term.

Increased postoperative pain, impaired balance reactions in the short, weak EMG responses of the trunk muscles, decreased pulmonary capacity and increased health costs have necessitated early rehabilitation in patients who had undergone scoliosis surgery. Also, the need for further research on the effects of physiotherapeutic approaches on the aforementioned functional losses has been indicated in several studies.Although early mobilization has been accepted as a rule of thumb by spinal surgeons in preventing the performance loss and reducing the causes of morbidity in recent years, the investigators could not find any research on postoperative rehabilitation implemented on patients under the supervision of a physiotherapist, following scoliosis surgery.

Therefore, based on these findings, the aim of this study was to compare effect of five days of intensive postoperative rehabilitation and mobilization on length of hospitalization and outcome in patients having scoliosis surgery.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of adolescent idiopathic scoliosis,
2. underwent posterior spinal fusion surgery,
3. Cobb's angle of 45 degrees or above,
4. were aged between 10 and 18 years.

Exclusion Criteria:

1. diagnosis of neuromuscular or rheumatismal diseases,
2. could not comply with the exercise program,
3. severe surgery-related pulmonary complications
4. complications which would prevent early rehabilitation (such as postoperative cerebrospinal fluid leak, paraparesis, hemiparesis),
5. surgery-related wound infections.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2017-02-05 (Actual); Primary Completion 2017-10-20 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
Pain via Visual Analogue Scale | Baseline, 1 week
  Change from baseline at 1 week Pain of the patients will be assessed by most widely used and accepted "visual analogue scale". It consists of a 10 centimeter line marked at one end with "no pain" and at other end with "worst pain ever". Patients is asked to indicate where on the line he or she rates the pain on the day of presentation, baseline, 1 week of follow-ups. Numerical score is given to it simply by measuring length between "no pain" to patients mark.
Thoracic Mobility Index | Baseline, 1 week
  Change from baseline at 1 week Thoracic mobility index was measured at the axillar, epigastric and subcostal regions during normal, maximal inspiration and maximal expiration, using a tape measure, baseline,1 week of follow-ups.

SECONDARY OUTCOMES:
Trunk Balance Test | Baseline, 1 week
  Change from baseline at 1 week Functional reach test was performed to assess the trunk balance. In standing position, the distances of sideways and forward reaches were measured as centimeters,baseline,1 week of followups.
2-minute Walking Test (2MWT) | Baseline, 1 week
  Change from baseline at 1 week Two-minute walking test (2MWT), the individual was asked to walk at normal pace for two minutes between the marked start and end points on a 30-meter-long corridor. The walking distance was measured in meters and recorded, baseline,1 week of followups.
Scoliosis Research Society-22 (SRS-22) | Baseline, 6 week
  Change from baseline at 1 week Scoliosis Research Society-22 (SRS-22) questionnaire was used to assess health-related quality of life. The questionnaire assesses pain, self-image, functions, mental health and satisfaction with the treatment. It consists of 22 items, each scored from 1, which is the worst situation, to 5, which is the best situation. The total score ranges from 1 to 5. Patients is asked to answer the questionnaire, baseline, 6 week of follow-ups.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Fatih Korkmaz, MD, Study Director — Inonu University Faculy of Medicine
Locations (1):
- Zilan Bazancir Apaydın, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: starting 12 months after publication
Access Criteria: Access criteria IPD and additional supporting information will share, analysis of primer and sekonder outcomes and clinical data will share after publication,

DOCUMENTS (2):
  • Informed Consent Form (2017-02-05): https://cdn.clinicaltrials.gov/large-docs/52/NCT04403152/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-02-05): https://cdn.clinicaltrials.gov/large-docs/52/NCT04403152/Prot_SAP_001.pdf